CLINICAL TRIAL: NCT07124416
Title: The Impact of the Adequacy of Keratinized Mucosa on Peri-implant Tissue Health and Patient-reported Outcomes
Status: Recruiting | Type: Observational
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-104
Record Dates: First submitted 2025-07-20; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- inadequate keratinized mucosa: peri-implant width of keratinized mucosa less than 2 mm
- adequate keratinized mucosa: peri-implant width of keratinized mucosa ≥ 2 mm
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention: observational case-control study
  Groups: adequate keratinized mucosa

SUMMARY:
This study aims to conduct a cross-sectional study to compare the differences in clinical indices, patient-reported outcomes, and levels of inflammatory factors in peri-implant gingival crevicular fluid between sites with adequate (≥ 2 mm) and inadequate (< 2 mm) keratinized mucosa after implant restoration, in order to explore the impact of the presence of keratinized mucosa on peri-implant soft and hard tissue health.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 70 years (inclusive of 18 and 70 years), of any gender;
* Patients who have undergone dental implant restoration是（single crown or fixed bridge restorations） at the Stomatology Hospital, Zhejiang University School of medicine and have had their final restoration for at least 6 months;
* Patients who voluntarily participate and sign the informed consent form after being fully informed, and who cooperate with relevant examinations.

Exclusion Criteria:

* Patients who are unwilling to participate in the follow-up of this study for various reasons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have completed dental implant restoration（single crown or fixed bridge restorations） for at least 6 months and undergo routine follow-up examinations.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Width of Keratinized Mucosa, KMW | on the day of enrollment
Plaque Index(PI) | on the day of enrollment
Bleeding on Probing(BOP) | on the day of enrollment
Peri-implant Probing Depth(PPD) | on the day of enrollment
Marginal Bone Loss(MBL) | The X-ray examination will be completed on the day of enrollment
Patient Satisfaction | on the day of enrollment
  visual analogue scale [VAS] 0-10,e.g., not at all satisfied to perfectly satisfied
Immunological parameters in peri-implant crevicular fluids(PICF) | The PICF will be collected on the day of enrollment
  PICF samples were collected from buccal aspects of implants after removing all supragingival plaque. The levels of IL-1β and PGE2 in PICF were measured using a sandwich ELISA kit.

CONTACTS AND LOCATIONS:
Locations (1):
- The Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China